CLINICAL TRIAL: NCT03785483
Title: Controlled Trial Testing the Effectiveness of Motivational Support on Physical Activity and Fatigue of Patients With Multiple Sclerosis
Brief Title: Implementation Intention for Physical Activity in Multiple Sclerosis
Acronym: apsep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: CeRSM (Unknown); COMUE (Unknown); Poissy-Saint Germain Hospital (Other); Hôpital Raymond Poincaré (Other); Paris West University Nanterre La Défense (Other); Cite Sep (Other)
Responsible Party: Principal Investigator, Ruffault Alexis, PhD, University of Paris 5 - Rene Descartes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: apsep-01
Record Dates: First submitted 2018-12-21; First posted 2018-12-24 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Motivation; Mindfulness
Keywords: Physical activity; Multiple sclerosis; Motivation; Intention; Mindfulness
MeSH Terms: conditions — Motor Activity; Multiple Sclerosis | interventions — Information Motivation Behavioral Skills Model; Mindfulness

STUDY DESIGN:
Intervention Model Description: 3 groups: motivation, mindfulness, and treatment as usual
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivation (Experimental): Using implementation intention techniques such as action planning. Every week, participants state when, where, and what kind of prescribed exercises they will do.
  Interventions: Behavioral: Motivation
- Mindfulness (Active Comparator): 10 minutes of audio recordings daily. Recordings contain: awareness of the breath, acceptation of thoughts and emotions, awareness of postures, awareness during stretching, awareness of a single movement (moving legs up while standing).
  Interventions: Behavioral: Motivation
- Treatment as usual (No Intervention): Physical activity prescribe 120 minutes per week.

INTERVENTIONS:
Behavioral: Motivation — 8 weeks of either action planning or mindfulness in addition to a treatment as usual which is a physical activity program of 120 minutes per week.
  Other Names: Mindfulness
  Arms: Mindfulness; Motivation

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an 8-week intervention based on implementation intention (motivation) in patients with multiple sclerosis on objectively measured physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged between 18 and 65 years
* Multiple sclerosis
* Recruited from CHU Poissy saint germain or Hôpital Raymond-Poincaré
* Informed consent provided during inclusion interview

Exclusion Criteria:

* Already participating in a clinical trial
* Cognitive dysfunctions in understanding simple guidelines
* Treatment reducing fatigue since less than 3 months
* Psychiatric disorders
* Unability to exercise
* Previous cardiovascular diseases
* Regular physical activity practice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-12-30 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity | From baseline to 3 months follow-up. Assessments at baseline, post-intervention (8 weeks), and 3 months follow-up.
  Accelerometer on a daily basis for 7 days

SECONDARY OUTCOMES:
Change in self-reported anxiety and depression (HADS) | From baseline to 3 months follow-up. Assessments at baseline, post-intervention (8 weeks), and 3 months follow-up.
  Hospital Anxiety and Depression Scale (2 subscales): anxiety (7 items) and depression (7 items) rated on a Likert-type scale ranging from 0 to 3. Total score for each subscale is the sum of each subscale's items. Higher scores indicate higher risks of anxiety and depression.
Change in self-reported mindfulness skills (FFMQ) | From baseline to 3 months follow-up. Assessments at baseline, post-intervention (8 weeks), and 3 months follow-up.
  Five-Facets Mindfulness Questionnaire (5 subscales): observing, describing, non-judging, non-reacting, acting with awareness. Each subscale is composed of 3 items rated on a Likert-type scale ranging from 1 to 5. Total score for each subscale is the sum of each subscale's items. Total mindfulness score is the sum of all subscales' scores. Higher scores indicate higher mindfulness skills.
Change in self-reported motivational regulation toward exercise (BREQ) | From baseline to 3 months follow-up. Assessments at baseline, post-intervention (8 weeks), and 3 months follow-up.
  Behavioral Regulation in Exercise Questionnaire (6 subscales): amotivation, external regulation, introjected regulation, integrated regulation, identified regulation, intrinsic regulation. Each subscale is composed of 3 items rated on a Likert-type scale ranging from 1 to 7. Total score for each subscale is the mean of each subscale's items. Higher scores indicate higher motivational regulation.
Change in self-reported beliefs toward physical activity (TPB). | From baseline to 3 months follow-up. Assessments at baseline, post-intervention (8 weeks), and 3 months follow-up.
  Theory of Planned Behavior constructs (4 concepts): attitudes (5 items), subjective norm (4 items), perceived behavioral control (2 items), intentions (3 items). All items are rated on a Likert-type scale ranging from 1 to 7. Total score for each subscale is the mean of each subscale's items. Higher scores indicate higher beliefs toward physical activity/

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Dematte, MSc, Principal Investigator — Paris Nanterre University
Locations (2):
- France (2):
  - Hôpital Raymond-Poincaré, Garches
  - CHU Poissy Saint germain, Poissy